CLINICAL TRIAL: NCT04921202
Title: First Affiliated Hospital of Jinzhou Medical Universtiy
Brief Title: Metabolic Syndrome and Degenerative Meniscus Lesions Related Knee Function
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Hongyu Wang, chief residents, The First People's Hospital of Jingzhou
Other Study IDs: Jinzhou Medical University
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Metabolic Syndrome; Meniscus Lesion; Obesity, Abdominal; Knee Arthritis
Keywords: Metabolic Syndrome; degenerate meniscus lesions; obesity; knee function
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- without metabolic syndrome and BMI<24: 100 volunteers aged between 35-70 years old with body mass index(BMI)<24 without Metabolic syndrome
- Metabolic Syndrome with BMI>27: 80 Metabolic syndrome patients with BMI>27 were included in the study
  Interventions: Other: Metabolic syndrome and meniscus injuries

INTERVENTIONS:
Other: Metabolic syndrome and meniscus injuries — Metabolic syndrome
  Groups: Metabolic Syndrome with BMI>27

SUMMARY:
Studies have suggested that Obese patients with metabolic syndrome(MetS)were correlated with knee joint degeneration and osteoarthritis. However, no studies demonstrate the relationship between obese patients with metabolic syndrome and degenerate meniscus lesions and its knee function.The aim is to detect the correlation between obese patients with metabolic syndrome and degenerate meniscus injuries.

DETAILED DESCRIPTION:
Obese patients with metabolic syndrome(MetS)were correlated with knee joint degeneration and osteoarthritis. However, no studies demonstrate the relationship between patients with metabolic syndrome and degenerate meniscus lesions or knee function. Participants were recruited from First Affiliated Hospital of Jinzhou Medical University. 100 BMI<24 people without Metabolic syndrome volunteers aged between 35-70 years old and 80 Metabolic syndrome patients with BMI>27 were included in the study. Obese patients with MetS were assessed knee function and degenerate meniscus tears verified by magnetic resonance imaging. And patients with a mild or no osteoarthritis with Kellgren and Lawrence grade<2 verified by X ray. We tested the relationship between metabolic syndrome and degenerate meniscus lesions. Obese patients with MetS and volunteers were detected by Mcmurry's test and MRI image to measure degeneration grade of meniscus tears. Number of MetS components were accounted and the knee function KOOS, IKDC score or degenerate meniscus tears were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 35 and 70 years old;
* Clinical diagnosis of metabolic syndrome;
* BMI score more than 27 or less than 24
* Clinical diagnosis of 3 grade degneration meniscus leisons;

Exclusion Criteria:

* Must be able to have no acute knee injury such as car crash or acute sports injury;
* Must be able to have no knee surgeries history;
* Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
* Must be able to have no contraindications to MRI;
* Must be able to have no severe cardiopulmonary disease;
* Must be able to have no musculoskeletal or neuromuscular impairments ;
* Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: participants from Jinzhou City, west of Liaoning Province
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
the Knee injury and Osteoarthritis Outcome Score (KOOS) total | up to 12 month
  The Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales including: Pain (9 items); other Symptoms (7 items); Activities of Daily Living (ADL, 17 items); Sport and Recreation function (Sport/Rec, 5 items); and knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems).
The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score | up to 12 month
  The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score to determine the meniscus function. The IKDC is a questionnaire that has high reliability and validity for patients with a meniscal tear[36, 37] [38]. The questionnaire contains 18 items (7 items for symptoms, 1 item for sport activity, 9 items for daily activities, and 1 item for current knee function.) The total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function and 0 is the worst.

SECONDARY OUTCOMES:
KOOS Pain subscale | up to 12 month
  Pain including 9 items，The minimum value is 0 and maximum values subscale is 100, the scored separately from zero (extreme knee problems) to 100 (no knee problems)
Symptoms subscale | up to 12 month
  Symptoms including 7 items,The minimum value is 0 and maximum values subscale is 100. Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
Activities of Daily Living subscale | up to 12 month
  Activities of Daily Living including 17 items,The minimum value is 0 and maximum values subscale is100. Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems).
Sport and Recreation function subscale | up to 12 month
  Sport and Recreation function including 5 items,The minimum value is 0 and maximum values subscale is 100. Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems).
knee-related Quality of Life subscale | up to 12 month
  knee-related Quality of Life including 4 items,The minimum value is 0 and maximum values subscale is 100. Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems).
KOOS4 | up to 12 month
  KOOS4, The minimum value is 0 and maximum values subscale is100. KOOS4 defined as the average score for four of the five knee injury and osteoarthritis outcome score (KOOS) validity for patients with meniscal tears and osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Wang, Doctor, Principal Investigator — The First People's Hospital of Jingzhou
Locations (1):
- First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided